CLINICAL TRIAL: NCT03903406
Title: Quality of Life, Symptoms and Treatment Satisfaction in Adult Patients With Relapsed and/or Refractory Multiple Myeloma, Receiving Ixazomib (Ninlaro®) in Combination With Lenalidomide and Dexamethasone in a Real World Setting: Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Multinational Center for Quality of Life Research, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: IISR-2018-102607
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
Keywords: quality of life
MeSH Terms: interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: ixazomib in combination with lenalidomide and dexamethasone — Patients with RRMM who have received at least one prior therapy will receive Ixazomib in combination with lenalidomide and dexamethasone within the routine clinical practice in accordance with prescription. Duration of therapy - until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this pilot study is to examine changes in patient-reported outcomes in patients with RRMM receiving triple therapy with ixazomib in combination with LenDex in a real world setting as well as to analyze clinical outcomes and safety of this treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with confirmed diagnosis of RRMM
* At least 18 years of age at the time of treatment start
* Patients who have received at least one prior therapy and who are suitable for treatment with ixazomib in combination with LenDex
* Patients who gave informed consent
* Patients who are capable to fill out questionnaires
* Patients with expected life duration of at least 6 months

Exclusion Criteria:

* Patients currently enrolled in any other clinical trials
* Patients with contraindications to ixazomib in accordance with instruction for use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with RRMM, who have received at least one prior therapy and who are suitable for triple therapy with ixazomib in combination with lenalidomide and dexamethasone. The eligibility criteria for this study are broader than the eligibility of patients to be treated with ixazomib in randomized clinical trials, so as to be reflective of routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Сhanges in quality of life (QoL) while treatment with ixazomib in combination with lenalidomide and dexamethasone as compared with baseline | Assessment of QoL changes will be done at 1, 3, 6, 9, 12 and 18 months after treatment with ixazomib in combination with lenalidomide and dexamethasone start as compared to baseline
  The change in QoL will be assessed as the difference in QoL means by scales of RAND SF-36 between any time-points during 18 mos of treatment and additionally as the difference in QoL means at any time-point as compared to baseline.
Changes in symptom severity while treatment with ixazomib in combination with lenalidomide and dexamethasone as compared with baseline | Assessment of changes in symptom severity will be done at 1, 3, 6, 9, 12 and 18 months after treatment with ixazomib in combination with lenalidomide and dexamethasone start
  The change in symptom severity will be assessed as the difference in the severity of each ESAS-R scale, the symptom distress score and the severity of NRS for assessing tingling hands/feet between any time-points during 18 mos of treatment and additionally at each time-point as compared with their baseline value. The proportion of patients with ≥1 point improvement on ESAS-R scale and on NRS for assessing tingling hands/feet at each time-point will be analyzed as well
Changes in number of satisfied/dissatisfied patients receiving ixazomib in combination with lenalidomide and dexamethasone | Assessment will be done at 1, 3, 6, 9, 12 and 18 months after treatment with ixazomib in combination with lenalidomide and dexamethasone start
  Changes in number of satisfied/dissatisfied patients receiving ixazomib in combination with lenalidomide and dexamethasone will be assessed at each time-point during treatment with ixazomib in combination with lenalidomide and dexamethasone

SECONDARY OUTCOMES:
Overall response rates and duration of response to treatment with ixazomib in combination with lenalidomide and dexamethasone | 18 mos from the start of treatment with ixazomib in combination with lenalidomide and dexamethasone
  Response to treatment will be assessed within the study and derived using the IMWG 2011 (International Myeloma Working Group). Duration of response will be evaluated from the time of initial response to treatment with ixazomib in combination with lenalidomide and dexamethasone till the disease progression or death from any cause
Progression free survival (PFS) in RRMM patients receiving ixazomib in combination with lenalidomide and dexamethasone | 18 mos from the start of treatment with ixazomib in combination with lenalidomide and dexamethasone
  PFS will be estimated from initiation of treatment with ixazomib in combination with lenalidomide and dexamethasone till the disease progression or death from any cause.
Overall survival (OS) in RRMM patients receiving ixazomib in combination with lenalidomide and dexamethasone | 18 mos from the start of treatment with ixazomib in combination with lenalidomide and dexamethasone
  OS will be estimated from initiation of treatment with ixazomib in combination with lenalidomide and dexamethasone till death from any cause
Frequency of adverse events (AEs)/serious AEs in RRMM patients receiving ixazomib in combination with lenalidomide and dexamethasone | 18 mos from the start of treatment with ixazomib in combination with lenalidomide and dexamethasone
  The analysis of safety of treatment with ixazomib in combination with lenalidomide and dexamethasone will include reporting adverse events (AEs)/serious AEs (SAEs). For adverse events assessment the NCI CTCAE v. 4.0 will be used. The incidence and severity of any AEs/SAEs will be evaluated within the study

IPD SHARING:
Plan to Share IPD: No